CLINICAL TRIAL: NCT00491062
Title: Analysis of Dopamine Neuronal Cell Loss Within the Enteric Nervous System in Parkinson's Disease
Brief Title: Enteric Nervous System in Parkinson's Disease
Acronym: ENTEROPARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Model: Parallel
Other Study IDs: 06-5-I
Record Dates: First submitted 2007-06-22; First posted 2007-06-25 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; enteric nervous system
MeSH Terms: conditions — Parkinson Disease | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Active Comparator)
  Interventions: Procedure: Biopsies
- Parkinson stade 1 (Experimental)
  Interventions: Procedure: Biopsies
- Parkinson stade2 (Experimental)
  Interventions: Procedure: Biopsies
- Parkinson stade 3 (Experimental)
  Interventions: Procedure: Biopsies

INTERVENTIONS:
Procedure: Biopsies

SUMMARY:
The "core" of the neuronal lesions in Parkinson's disease (PD) is the progressive degeneration of dopamine neurons in the substantia nigra. A significant loss of dopamine neurons and the presence of Lewy bodies (a pathological hallmark in PD) in enteric neurons have also been reported in that disease. These lesions may explain the frequent gastro-intestinal dysfunction observed in PD patients. Alterations of other neuronal populations within the enteric nervous system (ENS) as well as the mechanisms responsible for these lesions (type of cell death, alteration of neuromediators gene expression) remain to be identified. The aim of the study is to demonstrate that alterations of the human ENS in PD can be evidenced by bowel biopsies and to determine whether they are correlated to the severity of motor disability and to gastrointestinal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease patients at 3 different stages:

  * Early PD (before L-DOPA-induced complication);
  * Patients with L-DOPA-induced complication;
  * Patients with balance impairment or cognitive decline.
* Controls: patient at risk of colic cancer for whom a coloscopy is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-06; Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DAMIER Philippe, Study Director — Nantes University Hospital
Locations (1):
- CHU Nantes Gastro-enterologic and Neurologic Service, Nantes, Loire-Atlantique, France

REFERENCES:
- [Derived] Lebouvier T, Neunlist M, Bruley des Varannes S, Coron E, Drouard A, N'Guyen JM, Chaumette T, Tasselli M, Paillusson S, Flamand M, Galmiche JP, Damier P, Derkinderen P. Colonic biopsies to assess the neuropathology of Parkinson's disease and its relationship with symptoms. PLoS One. 2010 Sep 14;5(9):e12728. doi: 10.1371/journal.pone.0012728. PMID 20856865